CLINICAL TRIAL: NCT07295639
Title: Mobile Prenatal Education for Expectant Fathers and Its Effects on Bonding, Stress, Breastfeeding and Marital Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Sebahat Kuşlu, Research Assistant, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ethical Approval: 582.45.13
Record Dates: First submitted 2025-11-19; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breastfeeding Attitudes; Breast Feeding; Paternal Behavior; Health Education; Parent-Child Relations
Keywords: father-infant bonding; paternal stress; breastfeeding attitudes; mobile-based education
MeSH Terms: conditions — Breast Feeding; Health Education

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: an intervention group receiving mobile-based prenatal education for expectant fathers, and a control group receiving routine prenatal information. The outcomes of both groups will be compared after the intervention period.
Who Masked: Outcomes Assessor
Masking Description: This study is open-label for participants and investigators. However, the statistician responsible for data analysis will be blinded to group assignments to reduce potential bias in outcome evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-Based Prenatal Education for Expectant Fathers (Experimental): Fathers in this arm will receive access to a six-module mobile-based prenatal education programme covering infant care, nutrition and feeding, sleep routines, health and safety practices, emotional and social development, and daily care skills. They will complete pre- and post-intervention questionnaires on father-infant bonding, stress levels, and breastfeeding attitudes.
  Interventions: Behavioral: Mobile-based application
- Standard Routine Information for Expectant Fathers (No Intervention): Fathers in this arm will receive standard routine information provided in usual care. They will not have access to the mobile-based education programme. They will complete the same pre- and post-intervention questionnaires on father-infant bonding, stress levels, and breastfeeding attitudes during the same time intervals as the intervention group.

INTERVENTIONS:
Behavioral: Mobile-based application — The intervention is a six-module mobile-based training programme developed specifically for expectant fathers.
  The modules cover baby care, nutrition, sleep patterns, health and safety, emotional development and daily care.
  The aim is to strengthen the father-baby bond, reduce stress levels and develop a positive attitude towards breastfeeding.
  Arms: Mobile-Based Prenatal Education for Expectant Fathers

SUMMARY:
The aim of this interventional clinical trial is to assess whether a mobile-based antenatal education programme for expectant fathers has a positive effect on father-infant bonding, stress levels, and breastfeeding attitudes.

The study aims to answer the following main questions:

Does participation in a mobile-based prenatal education programme strengthen fathers' emotional bonds with their babies? Does the education reduce fathers' stress levels during the prenatal and postnatal periods? Does it increase the father's knowledge and supportive attitude towards breastfeeding? Researchers will compare whether there are measurable differences in attachment, stress, and breastfeeding attitudes between the intervention group (fathers receiving mobile-based education) and the control group (fathers receiving standard routine information).

Participants: Will complete pre- and post-intervention questionnaires assessing attachment, stress, and breastfeeding attitudes.

The intervention group will have access to a six-module mobile application covering topics such as infant care, nutrition, sleep routines, health and safety, emotional development, and daily care practices.

The study will be conducted with fathers aged 19-65 who became fathers within the last month and voluntarily agreed to participate.

DETAILED DESCRIPTION:
This interventional clinical trial aims to evaluate the effectiveness of a mobile-based prenatal education programme designed specifically for expectant fathers. The programme aims to strengthen father-infant bonding, reduce paternal stress levels during the prenatal and early postnatal periods, and enhance fathers' knowledge and supportive attitudes related to breastfeeding.

The study is grounded in the increasing scientific evidence demonstrating that fathers play an important role in maternal-infant health, emotional bonding, family cohesion, and early childhood development. Despite this, fathers frequently receive limited antenatal education and often feel unprepared for infant care, breastfeeding support, and the psychological transition to fatherhood. Mobile health (mHealth) technologies provide accessible, cost-effective, and father-friendly educational opportunities that help reduce participation barriers.

In this trial, participants will be randomly assigned to either an intervention group or a control group. Fathers in the intervention group will have access to a six-module mobile application that offers structured prenatal education. The modules cover infant care, nutrition and feeding, sleep routines, health and safety practices, emotional and social development, and daily care skills. The educational content is designed to support cognitive, emotional, and behavioural readiness for fatherhood and to enhance fathers' confidence in newborn care.

Participants in both groups will complete pre- and post-intervention questionnaires assessing father-infant bonding, stress levels, and breastfeeding attitudes. The intervention group will complete the post-test after engaging with the mobile application, while the control group will receive routine standard information and complete the same assessments during the same time periods. Differences between the two groups will be analysed to determine whether the mobile-based education leads to significant improvements in psychological and behavioural outcomes.

The study will be conducted with fathers aged 19-65 who have become fathers within the past month and who voluntarily agree to participate. Exclusion criteria include lack of smartphone access, inability to use mobile applications, or unwillingness to complete the questionnaires.

This trial is expected to contribute to the development of evidence-based perinatal care interventions that enhance paternal involvement within the domain of women's health nursing, support family-centred care models, and promote practices that strengthen maternal and infant health.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 65 years
* First-time father
* Has become a father within the last month
* Has a healthy newborn without congenital anomalies or chronic illnesses
* Does not have a premature or low-birth-weight baby
* Has not become a father through adoption
* Owns a mobile phone capable of accessing the mobile-based application
* Has an Android or iOS operating system
* Has not received any infant care training within the last 6 months
* Has no physical or mental disability that would prevent viewing, hearing, or understanding the research questions or educational content
* Voluntarily agrees to participate in the research

Exclusion Criteria:

* Declines to participate in the research
* Does not own a smartphone
* Cannot use mobile applications
* Has a physical or mental condition that prevents completing the questionnaires
* Has a baby with congenital anomalies or chronic medical conditions
* Has a premature or low-birth-weight baby
* Has received infant care training within the last 6 months
* Has adopted a child
* Is outside the 19-65 age range

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Paternal Stress Levels | Baseline (Day 1) and Post-Intervention (8 weeks after baseline)
  Paternal stress levels measured using the State-Trait Anxiety Inventory (STAI-State Subscale). A total score of 0-19 indicates no anxiety, a total score of 20-39 indicates mild anxiety, a total score of 40-59 indicates moderate anxiety, and a total score of 60-79 indicates severe anxiety. A total score of 60 or above indicates that the individual requires professional help.
Change in Father-Infant Bonding | Baseline (Day 1) and Post-Intervention (8 weeks after baseline)
  Father-infant bonding measured using the Father-Infant Bonding Scale. High scores on the scale indicate a high level of attachment.
Change in Breastfeeding Attitudes and Participation | Baseline (Day 1) and Post-Intervention (8 weeks after baseline)
  Fathers' attitudes and participation related to breastfeeding measured using the Fathers' Breastfeeding Attitude and Participation Scale. The total score under the sub-dimension of Fathers' Attitude Towards Breastfeeding ranges from 14 to 70, and the cut-off point for the scale is 58. The total score under the sub-dimension of Fathers' Participation in Breastfeeding ranges from 14 to 70, and the cut-off point for the scale is 58. High scores indicate high attitude and participation.
Change in Marital Satisfaction Levels | Baseline (Day 1) and Post-Intervention (8 weeks after baseline)
  Marital satisfaction measured using the Marital Satisfaction Scale. The total score that can be obtained from the scale, which consists of a single subscale, ranges from 12 to 60 points. There are no reverse items on the scale. An increase in the score obtained from the scale indicates a high level of marital satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Kuşlu, MSc, Principal Investigator — Gaziantep Islam Science and Technology University
Locations (1):
- Gaziantep Islam Science and Technology University, Şahinbey, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The ethics committee, confidentiality or national legislation deem sharing inappropriate.

REFERENCES:
- [Background] Bakker CJ, Wyatt TH, Breth MC, Gao G, Janeway LM, Lee MA, Martin CL, Tiase VL. Nurses' Roles in mHealth App Development: Scoping Review. JMIR Nurs. 2023 Oct 17;6:e46058. doi: 10.2196/46058. PMID 37847533
- [Background] Bich TH, Long TK, Hoa DP. Community-based father education intervention on breastfeeding practice-Results of a quasi-experimental study. Matern Child Nutr. 2019 Jan;15 Suppl 1(Suppl 1):e12705. doi: 10.1111/mcn.12705. PMID 30748110
- [Background] Challacombe FL, Pietikainen JT, Kiviruusu O, Saarenpaa-Heikkila O, Paunio T, Paavonen EJ. Paternal perinatal stress is associated with children's emotional problems at 2 years. J Child Psychol Psychiatry. 2023 Feb;64(2):277-288. doi: 10.1111/jcpp.13695. Epub 2022 Oct 10. PMID 36215991

DOCUMENTS (1):
  • Study Protocol (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT07295639/Prot_000.pdf